CLINICAL TRIAL: NCT03451214
Title: Effect of Zinc-Biofortified Wheat on Essential Fatty Acid Metabolism in Men
Brief Title: Evaluation of Zinc Intake on Essential Fatty Acid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHO22
Record Dates: First submitted 2018-02-09; First posted 2018-03-01 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-04

CONDITIONS: Inflammation; Oxidative Stress; Dyslipidemias
MeSH Terms: conditions — Inflammation; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diet zinc (Experimental): 3 dietary zinc levels: 6 mg/d, 11 mg/d and 25 mg supplemental zinc/d
  Interventions: Other: Diet Zinc

INTERVENTIONS:
Other: Diet Zinc — 4 mg zinc from zinc biofortified wheat, was added to a controlled diet; 25 mg supplemental zinc was given during the final recovery period

SUMMARY:
The purpose of this study is to determine the effect of different dietary zinc intakes on fatty acid metabolism and other zinc biomarkers

DETAILED DESCRIPTION:
This research is a dietary intervention study designed to evaluate the effect of progressive changes in Zn intake on fatty acid metabolism and to correlate those changes with biomarkers of dyslipidemia and insulin resistance. The main objective is to validate plasma fatty acid metabolism as a biomarker of inadequate Zn intake in subjects consuming identical diets with specific Zn content. The relative sensitivity of some fatty acid enzyme activities will also be compared to the DNA strand breaks. In addition to the primary objectives, correlations in enzyme activity with changes in fat metabolism, namely circulating triglyceride and cholesterol, will be determined. This will enable the determination of the effect of a low Zn intake on various aspects of dyslipidemia. Similar correlational analyses will be performed with clinical measures of inflammation and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* willing to limit food and beverage intake to that provided by the study
* willing to discontinue consumption of alcoholic beverages during the study
* willing to stop zinc supplementation 4 weeks prior to start of the study
* has an operative understanding of English
* no plans to move from the area during the study period

Exclusion Criteria:

* Chronic or acute metabolic disease
* smoker or user of nicotine products
* history of alcohol abuse, or use of illicit drugs.
* Is underweight or overweight, body mass index (BMI) < 18 or > 30 kg/m2.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Lipidomics changes | Day 0, day 15, day 57 and day 71
  Change in Fatty acid metabolism
DNA strand breaks changes | Day 0, day 15, day 57 and day 71
  change in COMET assay olive-tail moments

SECONDARY OUTCOMES:
Polar Metabolomics changes | Day 0, day 15, day 57 and day 71
  Change in Polar Metabolomics
Mineral analysis changes | Day 0, day 15, day 57 and day 71
  Changes in Plasma Zinc
Body weight changes | Day 0, day 15, day 57 and day 71
  changes in Body weight
Fat allocation changes | Day 0, day 15, day 57 and day 71
  Changes in waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Jung Suh, PhD, Principal Investigator — Associate Staff Scientist
Locations (1):
- UCSF Benioff Children's Hospital Oakland Research Institute, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liong EM, McDonald CM, Suh J, Westcott JL, Wong CP, Signorell C, King JC. Zinc-Biofortified Wheat Intake and Zinc Status Biomarkers in Men: Randomized Controlled Trial. J Nutr. 2021 Jul 1;151(7):1817-1823. doi: 10.1093/jn/nxab092. PMID 34036355